CLINICAL TRIAL: NCT06052709
Title: Investigation of Occupational Balance in Individuals With and Without Bruxism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 13.20
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Bruxism; Occupational Problems
Keywords: Bruxism; Occupational Balance; Stress
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with bruxism (Active Comparator): After the sociodemographic information of individuals is questioned, the presence and severity of temporomandibular joint disorders with the Fonseca Anamnestic Index, self-reported occupational balance with the Activity-Role Balance Questionnaire, and the individuals' stress levels with the Perceived Stress Scale will be evaluated.
  Interventions: Other: Occupational balance assessment
- Individuals without bruxism (Placebo Comparator): After the sociodemographic information of individuals is questioned, the presence and severity of temporomandibular joint disorders with the Fonseca Anamnestic Index, self-reported occupational balance with the Activity-Role Balance Questionnaire, and the individuals' stress levels with the Perceived Stress Scale will be evaluated.
  Interventions: Other: Occupational balance assessment

INTERVENTIONS:
Other: Occupational balance assessment — There is no intervention. The presence and severity of temporomandibular disorders, occupational balance, and stress levels of individuals will be evaluated.

SUMMARY:
Considering that occupational balance and bruxism are negatively affected by stress, this study aims to determine whether there is a difference in terms of occupational balance between individuals with and without bruxism.

DETAILED DESCRIPTION:
Occupation refers to daily life activities and task groups that are named, organized, given value and meaning by individuals and a culture. Occupation is everything people do to keep themselves busy, including taking care of themselves, enjoying life, and contributing to the social and economic fabric of their communities.

Bruxism is a parafunctional habit among temporomandibular disorders that occurs as a result of clenching and grinding teeth and overloading the stomatognathic structures. At the same time, bruxism is the chewing movement of the mandible, characterized by involuntary, rhythmic and non-functional teeth clenching and grinding, usually seen during sleep, and manifested by severe head and neck pain, limitation in jaw movements, pain and spasm in the chewing muscles. Although its etiology cannot be fully explained, it is thought that factors such as stress, occlusal disorders, allergies and sleep quality may be the source.

The deterioration or decrease in occupational balance may also be associated with people's quality of life. Occupational imbalance is reported to affect both physical and psychological state, creating significant stress on the body and mind, causing mental health problems and burnout.

Considering that occupational balance and bruxism are negatively affected by stress, this study aims to determine whether there is a difference in terms of occupational balance between individuals with and without bruxism.

ELIGIBILITY:
Inclusion Criteria:

* To be volunteer

Exclusion Criteria:

* Psychological disorders,
* Neurological disorders,
* Orthopedic disorders,
* Cognitive impairment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Fonseca Anamnestic Index | up to 3 months
  The presence and severity of temporomandibular disorders in individuals will be questioned with the Fonseca Anamnestic Index. The Fonseca Anamnestic Index consists of 10 questions. The participant is asked to answer each question as 'Yes' (10 points), 'No' (0 points), and 'Sometimes' (5 points). The questionnaire score is given points for all questions, and the severity of temporomandibular disorders is classified according to the total score: no temporomandibular disorders (0-15 points), mild temporomandibular disorders (20-40 points), moderate temporomandibular disorders (45-65 points), severe temporomandibular disorders (70-100). Turkish version, validity, and reliability study was conducted.
Occupational Balance Questionnaire | up to 3 months
  Occupational Balance Questionnaire is a scale that measures self-reported occupational balance in different dimensions. The purpose of the scale is to measure the satisfaction of the individual according to the amount and variety of daily activities and to define his/her occupational balance according to the results obtained. The 11 items in the scale are scored on a 4-point scale from "strongly disagree" to "strongly agree". The total score is obtained by summing the individual items and ranges from 0 to 33, with higher scores indicating greater occupational balance. Turkish version, validity and reliability study was conducted.
Perceived Stress Scale | up to 3 months
  Individuals' stress levels will be measured with the Perceived Stress Scale. The Perceived Stress Scale, consisting of 14 items, measures how stressful some situations in a person's life are perceived. Participants evaluate each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". 7 of the items containing positive statements are reverse scored-scores of the Perceived Stress Scale range from 0 to 56. A high score indicates a person's perception of stress is high. A Turkish version, validity, and reliability study of the Perceived Stress Scale was conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)